CLINICAL TRIAL: NCT00634166
Title: Prospective Evaluation of the Effects of Topical Therapy With Sulfamylon® For 5% Topical Solution on Autograft Healing in Subjects With Thermal Injuries Requiring Meshed Autografts: A Comparison to a Historical Control Group
Brief Title: Effects of Therapy With Sulfamylon® 5% Topical Solution Compared to a Historical Control Group
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA request as study could not serve as the confirmatory trial.
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan Bertek Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMS-401
Record Dates: First submitted 2008-02-11; First posted 2008-03-12 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Burns
Keywords: thermal injuries; burns; Burn Patients
MeSH Terms: conditions — Burns | interventions — Mafenide; Solutions; Anti-Infective Agents; Bacitracin; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Historical Control (Other): Treated within the last 5 years (if possible) with topical prophylactic therapies that did not include mafenide acetate or mafenide salt forms. These are considered the Topical Antimicrobial/Antifungal Medications
  Interventions: Drug: Topical Antimicrobial/Antifungal Medications
- Prospective Patients/Active Drug (Experimental): Prospective subjects with thermal injuries of 20-60% TBSA on the chest, abdomen, or proximal upper and lower extremities requiring meshed autografts on these areas will receive SS5% as the initial topical moist dressing over the meshed autograft(s) placed at the initial graft procedure (Day 1). Intervention is Sulfamylon® For 5 % Topical Solution.
  Interventions: Drug: Sulfamylon® For 5 % Topical Solution

INTERVENTIONS:
Drug: Sulfamylon® For 5 % Topical Solution — Sulfamylon® For 5% Topical Solution is indicated for use as an adjunctive topical antimicrobial agent to control bacterial infection when used under moist dressings over meshed autografts on excised burn wounds.
  Other Names: mafenide acetate
  Arms: Prospective Patients/Active Drug
Drug: Topical Antimicrobial/Antifungal Medications — 'Topical Antimicrobial/Antifungal Medications' Various topical antimicrobials and antifungals include: Bacitracin; Amphotericin B; Silver Sulfadiazine; Cefazolin; Vancomycin; Nystatin; Fluconazole; Piperacillin Sodium with Tazobactam.
  Other Names: Bacitracin; Amphotericin B; others noted below.
  Arms: Historical Control

SUMMARY:
The primary objective is to compare the effectiveness of treatment with Sulfamylon® solution as the initial topical moist dressing over meshed autografts following the initial graft procedure on preventing graft loss in a prospective cohort of subjects versus a historical control group in a non-inferiority trial.

DETAILED DESCRIPTION:
This is a prospective, non-inferiority, multi-center, historically controlled, open label study that will evaluate the effects of topical therapy with Sulfamylon® For 5% Topical Solution on autograft healing in subjects with thermal injuries requiring meshed autografts against a similar historic control population in which Sulfamylon® For 5% Topical Solution or mafenide acetate or other mafenide salt forms were not used. Prospective subjects meeting the entrance criteria will receive Sulfamylon® solution as topical antimicrobial treatment on moist dressings following initial meshed autograft procedure (Day 1). Sulfamylon® solution will be used every 6-8 hours, or as needed, to keep the dressing moist. The graft will be evaluated on Days 5-7, Days 12-14 and Days 18-21, unless the subject is discharged, dies, or experiences graft loss / regrafting of the initial meshed autograft prior to Assessment 4 (Days 18-21).

ELIGIBILITY:
Inclusion Criteria:

In order for prospective subjects to be eligible for entry into the study:

* Subjects must have thermal injuries of 20-60% TBSA requiring at least one meshed autograft on the chest, abdomen, or proximal upper and lower extremities following surgical excision of the burn injury. Refer to Supplement 20.3.2: Lund Browder charts
* Subjects may be male or female, 3 months of age or older
* Females of childbearing potential must have a negative urine pregnancy test upon admission and agree to avoid pregnancy throughout the course of the study. Since this population is hospitalized for the duration of the study, an agreement of sexual abstinence is appropriate for this trial. Those subjects who do not wish to commit to sexual abstinence for the duration of this study must agree to avoid pregnancy by using a medically supervised method of contraception (such as hormonal contraception in conjunction with a vaginal spermicide or a tubal ligation at least 3 months prior to study entry)
* Subjects must be willing and able to provide written informed consent. If subjects are unable to provide written informed consent, then the subject's legally acceptable representative may provide written informed consent in accordance with the IRB/IEC, and federal, state and local regulations.

Exclusion Criteria:

Prospective subjects will be excluded from the study for the following reasons:

* Non-thermal burn injuries
* Inhalation injuries resulting in a PaO2 /FIO2 ratio < 300 mmHg on more than one arterial blood gas in the first 48 hours post-admission
* Females who are currently pregnant or breast feeding, or who intend to become pregnant during the course of the study
* Subjects with acute renal failure
* Subjects with known systemic allergy to sulfonamides or to sulfur-containing medication
* Time interval between burn injury and excision and grafting is greater than 7 days
* Grafting procedures that are conducted and/or evaluated on an outpatient basis
* Inability to use a meshed autograft as part of the initial grafting procedure
* Inability to use SS5% as the only initial prophylactic topical antimicrobial therapy on meshed autografts
* Thermal burn injuries less than 20% or greater than 60% TBSA
* Subjects who are participating in any other clinical studies involving any investigational product, or who have participated in such a study within the previous 30 days
* Subjects with known glucose-6-phosphate dehydrogenase deficiency

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Davis, MD, Study Director — Mylan Inc.
Locations (9):
- United States (9):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Arrowhead Regional Medical Center, Redlands, California
  - Shands Burn Center - Univ. of Florida, Gainesville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - The Plastic Surgery Institute - Southern Illinois Univ. School of Medicine, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - John's Hopkins Burn Center, Baltimore, Maryland
  - University of Missouri Healthcare - Dept. of Surgery, Columbia, Missouri
  - Wake Forest University - Department of General Surgery, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Control: Treated within the last 5 years (if possible) with topical prophylactic therapies that did not include mafenide acetate or mafenide salt forms (with the sponsor's prior approval, sites may obtain historical control subjects treated longer than 5 years ago)
  Sulfamylon® (mafenide acetate) For 5 % Topical Solution: Sulfamylon® For 5% Topical Solution is indicated for use as an adjunctive topical antimicrobial agent to control bacterial infection when used under moist dressings over meshed autografts on excised burn wounds.
- Prospective Patients/Active Drug: Prospective subjects with thermal injuries of 20-60% TBSA on the chest, abdomen, or proximal upper and lower extremities requiring meshed autografts on these areas will receive SS5% as the initial topical moist dressing over the meshed autograft(s) placed at the initial graft procedure (Day 1).
  Sulfamylon® (mafenide acetate) For 5 % Topical Solution: Sulfamylon® For 5% Topical Solution is indicated for use as an adjunctive topical antimicrobial agent to control bacterial infection when used under moist dressings over meshed autografts on excised burn wounds.
Period: Overall Study
Arm/Group | Historical Control | Prospective Patients/Active Drug
Started | 82 | 138
Completed | 22 | 78
Not Completed | 60 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Control | Prospective Patients/Active Drug | Total
Number analyzed (Participants) | 82 | 138 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (18.91) | 44.7 (17.87) | 42.6 (18.44)
Age, Customized [Number; unit: participants]
  <18 years | 11 | 5 | 16
  >= 18 years | 71 | 133 | 204
Sex/Gender, Customized [Number; unit: participants]
  Female | 19 | 29 | 48
  Male | 63 | 109 | 172
Region of Enrollment [Number; unit: participants]
  United States | 82 | 138 | 220

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Graft Loss After Initial Meshed Autograft Procedure on Days 5-7.
Time Frame: The primary analysis will compare the percent of subjects with All Cause Graft Loss of the initial meshed autograft procedure at Days 5-7.
Measure: Number; unit: Percentage of Participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of Participants | 4.9 | 4.3

2. Secondary Outcome: Percentage of Participants With All-cause Graft Loss at Days 12 to 14 in the FAS Population
Description: All cause graft loss is defined as graft adhesion of < 85% for the initial meshed autograft procedure.
Time Frame: Secondary analyses will include the percent of subjects with All Cause Graft Loss at Days 12-14
Measure: Number; unit: Percentage of participants
Groups:
- Historical Control: .Treated within the last 5 years (if possible) with topical prophylactic therapies that did not include mafenide acetate or mafenide salt forms (with the sponsor's prior approval, sites may obtain historical control subjects treated longer than 5 years ago) Sulfamylon® (mafenide acetate) For 5 % Topical Solution: Sulfamylon® For 5% Topical Solution is indicated for use as an adjunctive topical antimicrobial agent to control bacterial infection when used under moist dressings over meshed autografts on excised burn wounds.
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 20.3 | 2.7

3. Secondary Outcome: Percentage of Participants With All-cause Graft Loss at Days 18 to 21 in the FAS Population
Description: All cause graft loss is defined as graft adhesion of < 85% for the initial meshed autograft procedure.
Time Frame: Days 18 to 21
Measure: Number; unit: Percentage of participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 4.5 | 6

4. Secondary Outcome: Percentage of Participants With Treatment Failure at Days 5 to 7 in the FAS Population
Description: Treatment failure is defined as a change in topical antimicrobial therapy of initial meshed autograft due to suspected infection within the first 7 days or infectious graft loss.
Time Frame: Days 5-7
Measure: Number; unit: Percentage of participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 13.4 | 1.4

5. Secondary Outcome: Percentage of Participants With Infectious Graft Loss at Days 5 to 7 in the FAS Population
Description: Graft adhesion of < 85% for the initial meshed autograft procedure due to infection.
Time Frame: Days 5-7
Measure: Number; unit: Percentage of participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 2.4 | 0.7

6. Secondary Outcome: Percentage of Participants With Infectious Graft Loss at Days 12 to 14 in the FAS Population
Description: Graft adhesion of < 85% for the initial meshed autograft procedure due to infection.
Time Frame: Days 12-14
Measure: Number; unit: Percentage of participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 3.4 | 0.0

7. Secondary Outcome: Percentage of Participants With Infectious Graft Loss at Days 18 to 21 in the FAS Population
Description: Graft adhesion of < 85% for the initial meshed autograft procedure due to infection.
Time Frame: Days 18-21
Measure: Number; unit: Percentage of participants
Arm/Group | Historical Control | Prospective Patients/Active Drug
Number analyzed (Participants) | 82 | 138
Percentage of participants | 0.0 | 1.3

ADVERSE EVENTS:
Description: There is a change in the analysis sets that were used for analyzing efficacy-FA Set and Safety data- Safety set. Out of 138 patients enrolled, one patient had 'No post-graft assessments' and hence the patient was excluded from FAS- efficacy analysis. This resulted in a reduced number(one less) of patients for FAS. There is no analytical error.
  Reference -Table 14.1.3.1
Arm/Group | Historical Control | Prospective Patients/Active Drug
Serious Adverse Events (participants affected / at risk) | 9/82 | 27/138
Other Adverse Events (participants affected / at risk) | 74/82 | 130/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Historical Control (N=82) | Prospective Patients/Active Drug (N=138)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Multi-organ Failure (General disorders) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5)
Sepsis (Infections and infestations) | 2 (2) | 9 (12)
Renal Failure (Renal and urinary disorders) | 1 (1) | 6 (6)
Renal Failure - acute (Renal and urinary disorders) | 2 (2) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 9 (9)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Historical Control (N=82) | Prospective Patients/Active Drug (N=138)
Anaemia (Blood and lymphatic system disorders) | 16 (20) | 27 (30)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 12 (12)
Thrombocythaemia (Blood and lymphatic system disorders) | 7 (8) | 14 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 7 (7)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 9 (9)
Tachycardia (Cardiac disorders) | 4 (4) | 20 (20)
Constipation (Gastrointestinal disorders) | 34 (42) | 42 (48)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 10 (11)
Nausea (Gastrointestinal disorders) | 13 (13) | 18 (18)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (8)
Pyrexia (General disorders) | 12 (13) | 20 (35)
Bacteraemia (Infections and infestations) | 2 (2) | 10 (10)
Cellulitis (Infections and infestations) | 3 (3) | 7 (7)
Pneumonia (Infections and infestations) | 16 (17) | 19 (22)
Sepsis (Infections and infestations) | 3 (3) | 11 (14)
Urinary Tract Infection (Infections and infestations) | 7 (7) | 11 (13)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 8 (17)
Procedural Pain (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Culture Wound Positive (Investigations) | 5 (12) | 5 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 17 (17)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 10 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (7) | 9 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (12) | 13 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 13 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (8) | 16 (17)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 7 (8)
Agitation (Psychiatric disorders) | 8 (8) | 19 (19)
Anxiety (Psychiatric disorders) | 7 (7) | 15 (16)
Depression (Psychiatric disorders) | 3 (3) | 8 (8)
Insomnia (Psychiatric disorders) | 12 (12) | 23 (26)
Renal Failure (Renal and urinary disorders) | 2 (2) | 8 (8)
Renal Failure-acute (Renal and urinary disorders) | 3 (3) | 9 (9)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13) | 25 (28)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 9 (9)
Hypertension (Vascular disorders) | 4 (4) | 13 (13)
Hypotension (Vascular disorders) | 5 (5) | 13 (27)

LIMITATIONS AND CAVEATS:
The study was terminated on 17 June 2013 due to the recommendation and request by the FDA to design a superiority clinical study to satisfy the sponsor's post marketing study commitment for SS5%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall provide Sponsor with (i) a copy of the papers prepared for publication by him or her as soon as possible, but in any event not less than sixty (60) days prior to their submission to a scientific journal or other publication; or (ii) a reasonably detailed summary or abstract of any oral presentation not less than forty-five (45) days prior to their submission or presentation. Sponsor may comment and remove any confidential information as needed.